CLINICAL TRIAL: NCT05058352
Title: A Phase I, Open-label，Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS269, in Patients With Advanced Solid Tumor
Brief Title: A Study of HS269 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS269-Ⅰ-01
Record Dates: First submitted 2021-09-02; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS269 (Experimental): Multiple doses of HS269 tablets
  Interventions: Drug: HS269

INTERVENTIONS:
Drug: HS269 — Oral tablets, once daily. Dose escalation from 50 mg QD, through 100 mg, 200mg, 300 mg, 400 mg, to 500mg.

SUMMARY:
This is a Phase I, open-label, first in human study of HS269 tablet, a small molecule highly-selective RET Inhibitor. The dose-escalation study will assess the safety, tolerability, and pharmacokinetics of HS269 and determine the dose and schedule to be used in Phase II. Seventeen to thirty-six patients with advanced solid tumor may be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years, no gender limit.
2. Patients with advanced solid tumors confirmed by histology or cytology fail to receive standard treatment, or there is no standard treatment, or standard treatment is not applicable at this stage.
3. At least one evaluable tumor lesion according to RECIST version 1.1.
4. ECOG≤ 1.
5. The estimated survival time was more than 3 months.
6. The function of all organs was good, the specific indexes were as follows:

   Blood system (no transfusion or hematopoietic stimulating factor treatment within 14 days) i. #NEUT ≥1.5×109/L ii. PLT ≥90×109/L iii. HGB ≥85g/L Liver function i. TBIL ≤1.5×ULN ii. ALT ≤3×ULN; Patients with liver metastasis or liver cancer: ≤ 5 × ULN iii. AST ≤3×ULN; Patients with liver metastasis or liver cancer: ≤ 5 × ULN Renal function i. Ccr >50 ml/min（According to Cockcroft-Gault formula） Blood coagulation function i. APTT ≤1.5×ULN ii. INR ≤1.5×ULN
7. The subjects should be informed and agreed to the study before the start of the trial, and sign the written informed consent voluntarily.

Exclusion Criteria:

1. Received anti-tumor treatments within 14 days or less than 5 half-lives (whichever is longer) before the first use of the study drug
2. Received blood transfusion, erythropoietin, recombinant human thrombopoietin or colony stimulating factor and other treatments within 7 days before receiving blood system examination during the screening period.
3. Received other unmarketed clinical study drugs or treatments within 4 weeks before the first use of the study drug.
4. Major organ surgery (excluding biopsy) or significant trauma occurred within 4 weeks before the first use of the study drug;
5. Systemic administration of glucocorticoids (prednisone > 10 mg / day or equivalent dose of the same drug) or other immunosuppressants within 14 days before the first use of the study drug; except for local, eye, intra articular, nasal and inhaled corticosteroids; short-term use of glucocorticoids for preventive treatment (e.g. prevention of contrast agent allergy)；
6. CYP1A2/P-gp potent inhibitors or potent inducers were used within 7 days before the first use of the study drug；
7. Resistance to selective RET inhibitors;
8. The adverse reactions of previous anti-tumor therapy have not yet recovered to CTCAE 5.0 grade evaluation ≤ 1 (except for the toxicity without safety risk judged by researchers such as alopecia)；
9. Patients with central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence indicating that the central nervous system metastasis or meningeal metastasis has not been controlled, which is not suitable for the study.
10. Have active infection and need systemic anti infection therapy；
11. Have a history of immunodeficiency, including HIV antibody test positive；
12. Active hepatitis B, allowing preventive antiviral treatment other than interferon; hepatitis C virus infection；
13. Present or past interstitial lung disease (except radiation-induced pulmonary fibrosis without hormone therapy)；
14. Poorly controlled diabetic patients.
15. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. Serious abnormal cardiac rhythm or conduction, such as ventricular arrhythmia, Ⅱ - Ⅲ degree atrioventricular block, etc;
    2. In the resting state, average QTcF≥480ms in 12 lead -ECG；
    3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular events of grade 3 or above occurred within 6 months before the first administration;
    4. NYHA ≥II or LVEF<50％；
    5. Hypertension beyond clinical control；
16. Could not take medication orally，or have severe gastrointestinal obstruction (such as gastrointestinal obstruction, gastrointestinal absorption)；
17. The third space effusion, which could not be controlled clinically, was not suitable for the study；
18. Mental disorder or poor compliance；
19. Eligible patients with fertility (male and female) do not agree to use reliable contraceptive methods (abstinence, condom, intrauterine device or ligation) with their partner during the trial and for at least 3 months after the last medication.
20. Female patients have a positive blood pregnancy test within 7 days before enrollment, or breastfeeding women;
21. The subjects were not suitable for the clinical study because of other serious systemic diseases or other reasons according to the investigator 's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | From date of initial dose until up to 33 days for treatment
  Incidence rate of dose limiting toxicities (DLT)
Adverse Event(s) and Serious Adverse Event(s) | Through study completion or early study discontinuation（up to 12 months）
  The occurrence and rate of AE and SAE

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | From date of initial dose until up to 33 days for treatment
  Cmax of HS269
Area Under the Plasma Concentration versus Time Curve (AUC) | From date of initial dose until up to 33 days for treatment
  AUC of HS269
Calcitonin in Peripheral Blood | Through study completion or early study discontinuation（up to 12 months）
  For Medullary Thyroid Cancer patients
Thyroglobulin in Peripheral Blood | Through study completion or early study discontinuation（up to 12 months）
  For non-MTC thyroid cancer patients
ORR | Approximately 12 months
  Objective response rate (ORR)
DCR | Approximately 12 months
  Disease control rate (DCR)
PFS | Approximately 12 months
  Progression free survival (PFS)
Peripheral blood ctDNA | Through study completion or early study discontinuation（up to 12 months）
  Only for patients with positive RET gene mutation

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Principal Investigator — Henan Provincial People's Hospital; Qi Dang, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided